CLINICAL TRIAL: NCT04422340
Title: A Multicentric Survey on Patients Over 60 Admitted to Intensive Care for Severe Forms of COVID Infection: Search for Prognostic Criteria Associated With Survival
Brief Title: Senior-COVID-Rea Multicentric Survey
Acronym: SeniorCOVIDRea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0386
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: COVID-19 Disease, Severe Form

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Group1 — * Comorbidities (CIRS-G scale),
  * Functional status of the patient with
    * Clinical frailty scale (1 month before infection)
    * ADL score (1 month before infection)
  * Biological data
    * Blood group
    * TP, D-dimers, CRP, creatinine level at the patient's entry, triglyceridemia, fibrinogen, ferritin
    * Parameters derived from the platelet formula count on D1 of the start of intensive care (lymphocytes, neutrophils, platelets, average platelet volume, red blood cell distribution index), SYSMEX data (IG: Immature granulocytes; HFLC: high fluorescent lymphocyte count)
  * Resuscitation outcomes
    * LDH rate at the start of intensive care
    * PaO2 / FiO2 ratio at the start of intensive care
    * IGSII / SASPII score (simplified acute physiology score) on D1 of the start of intensive care
    * SOFA score (sepsis-related organ failure assessment): a posteriori estimate based on IGSII / SASPII
    * Delay between the appearance of the first signs of infection and admission to intensive care

SUMMARY:
With the spread of COVID-19 epidemic since 2019 in Wuhan, China health plans have to be adapted continuously in response to the emergency. The first publications from the Chinese experience demonstrate an increase in the incidence of COVID-19 infections in patients over 60 years of age, a higher frequency of severe forms of the disease and therefore theoretical indications of orientation towards resuscitative care.

However, the first published data from Hubei province suggest a low benefit of resuscitation for patients between 70 and 80 years of age and null in patients over 80 years of age. These data question the individual benefit / risk balance of an orientation towards resuscitation for this category of patients, their quality of life and the concept of unreasonable obstinacy.

Among the covariates associated with resuscitation mortality described in the data published to date, cardiovascular comorbidities, certain biological covariates (LDH, creatinine, lymphocytes, neutrophils, TP, D-dimers, etc.), the time between the first symptoms and the entry into resuscitation have been identified.

The objective of this multicentric observational study is to determine the clinical and biological covariates predictive of mortality in the population of patients over 60 years of age admitted in intensive care unit, in particular by integrating functional and nutritional data from patients 1 month before COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 60
* sent to the intensive care unit
* whose COVID diagnosis has been established (RT-PCR and / or chest scanner)

Exclusion Criteria:

* Refusal of the patient or his support person to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 60 in intensive care unit for severe COVID infection
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of age on mortality at 30 days after admission to intensive care | 30 days after resuscitation admission
  First hypothesis: considering a single analysis variable (age), with expected mortality of 30% in patients under 70, and 70% in patients over 70 (with 40% of patients over 70), a total of 130 patients is necessary to show a statistically significant difference between these two groups with a power of 90% (bilateral alpha risk test of 5%). Since the multivariate analysis considers the integration of several factors, considering 15 factors, hoping for a coefficient of determination of 0.5 of the model, to achieve an optimism of less than 10%, it will be necessary to include 185 patients.
  After the publication of data on mortality in ICU in Lombardy region, Italy in April 2020, it was considered that a stopping of the trial at 185 patients would impair its statistical power and induce a potential risk of patients' selection bias. As a consequence the scientific committee decided that all the patients admitted to ICU until May 7th would be proposed the study.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Falandry, MD, Principal Investigator — Hospices Civils de Lyon
Locations (7):
- France (7):
  - Resuscitation unit at Hospital Emile Roux, Le Puy-en-Velay
  - - Resuscitation unit of the Groupement Hospitalier Nord - Hospices Civils de Lyon, Lyon
  - - Resuscitation unit of the Groupement Hospitalier Sud - Hospices Civils de Lyon, Lyon
  - Resuscitation unit of the Groupement Hospitalier Centre - Hospices Civils de Lyon, Lyon
  - Resuscitation unit of the Groupement Hospitalier Sud - Hospices Civils de Lyon, Lyon
  - Service de Réanimation de l'Hôpital Nord Ouest, Villefranche-sur-Saône
  - Medipole Resuscitation unit, Villeurbanne

REFERENCES:
- [Derived] Thiolliere F, Falandry C, Allaouchiche B, Geoffray V, Bitker L, Reignier J, Abraham P, Malaquin S, Balanca B, Boyer H, Seguin P, Guichon C, Simon M, Friggeri A, Vacheron CH; AZUREA Study Group. Intensive care-related loss of quality of life and autonomy at 6 months post-discharge: Does COVID-19 really make things worse? Crit Care. 2022 Apr 4;26(1):94. doi: 10.1186/s13054-022-03958-6. PMID 35379312
- [Derived] Falandry C, Malapert A, Roche M, Subtil F, Berthiller J, Boin C, Dubreuil J, Ravot C, Bitker L, Abraham P, Collange V, Balanca B, Goutte S, Guichon C, Gadea E, Argaud L, Dayde D, Jallades L, Lepape A, Pialat JB, Friggeri A, Thiolliere F; Senior-COVID-Rea study Group. Risk factors associated with day-30 mortality in patients over 60 years old admitted in ICU for severe COVID-19: the Senior-COVID-Rea Multicentre Survey protocol. BMJ Open. 2021 Jul 6;11(7):e044449. doi: 10.1136/bmjopen-2020-044449. PMID 34230013